CLINICAL TRIAL: NCT06866951
Title: CIT Trial for Cervical Cancer Patients
Brief Title: A Clinical Study Comparing Chemotherapy Combined With PD-1 Inhibitor Versus Concurrent Chemoradiotherapy in Cervical Cancer Patients With Positive Lymph Nodes After Surgery: A Multicenter Randomized Controlled Clinical Trial
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO2024-777
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Cervical Cancers
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemo-immunotherapy group (Experimental): Post-radical surgery for cervical cancer, the first cycle of PD-1 inhibitor combined with chemotherapy will begin 2 to 3 weeks after surgery. Each treatment cycle lasts 21 days, with a total of 6 cycles. A complete imaging efficacy evaluation will be conducted after every 3 treatment cycles. For patients with lymph node metastasis ≥3 or para-aortic lymph node metastasis, 6 cycles of chemotherapy combined with immunotherapy will be administered. Other patients will receive 3 cycles of chemotherapy combined with immunotherapy.
  Treatment regimen:
  Day 1:
  Paclitaxel (albumin-bound) for injection: 260 mg/m², administered intravenously over 30 minutes.
  Day 1 to Day 2:
  Cisplatin 75-80 mg/m², administered intravenously at a 1 mg/min rate.
  Day 3:
  PD-1 inhibitor (Camrelizumab for injection, Aikening): 200 mg per dose, infused over 30 to 60 minutes.
  Interventions: Drug: Chemo-immunotherapy
- CCRT group (Active Comparator): Standard treatment includes cisplatin, external beam radiotherapy (EBRT), and brachytherapy.
  The overall chemoradiotherapy (including EBRT and brachytherapy) should typically be completed within 6 weeks (with a maximum extension to 10 weeks in case of anticipated delays). External beam radiotherapy (EBRT) should be at least three-dimensional conformal radiotherapy, with image-guided (CT or MR) intensity-modulated conformal radiotherapy techniques recommended, at a 45-50 Gy dose.
  Concurrent Chemotherapy:
  Cisplatin (40 mg/m²) is preferred on a weekly schedule (administered before the planned EBRT on the same day, once a week [±1-day window], for a total of 5-6 infusions). Carboplatin can be used as an alternative if cisplatin toxicity is not tolerated.
  Interventions: Radiation: CCRT

INTERVENTIONS:
Drug: Chemo-immunotherapy — Post-radical surgery for cervical cancer, the first cycle of PD-1 inhibitor combined with chemotherapy will begin 2 to 3 weeks after surgery. Each treatment cycle lasts 21 days, with a total of 6 cycles. A complete imaging efficacy evaluation will be conducted after every 3 treatment cycles. For patients with lymph node metastasis ≥3 or para-aortic lymph node metastasis, 6 cycles of chemotherapy combined with immunotherapy will be administered. Other patients will receive 3 cycles of chemotherapy combined with immunotherapy.
  Treatment regimen:
  Day 1:
  Paclitaxel (albumin-bound) for injection: 260 mg/m², administered intravenously over 30 minutes.
  Day 1 to Day 2:
  Cisplatin 75-80 mg/m², administered intravenously at a 1 mg/min rate.
  Day 3:
  PD-1 inhibitor (Camrelizumab for injection, Aikening): 200 mg per dose, infused over 30 to 60 minutes.
  Arms: Chemo-immunotherapy group
Radiation: CCRT — The overall chemoradiotherapy (including EBRT and brachytherapy) should typically be completed within 6 weeks (with a maximum extension to 10 weeks in case of anticipated delays). External beam radiotherapy (EBRT) should be at least three-dimensional conformal radiotherapy, with image-guided (CT or MR) intensity-modulated conformal radiotherapy techniques recommended, at a 45-50 Gy dose.
  Concurrent Chemotherapy:
  Cisplatin (40 mg/m²) is preferred on a weekly schedule (administered before the planned EBRT on the same day, once a week [±1-day window], for a total of 5-6 infusions). Carboplatin can be used as an alternative if cisplatin toxicity is not tolerated.
  Arms: CCRT group

SUMMARY:
This study aims to conduct a prospective, multicenter, randomized controlled trial targeting patients with cervical cancer who have been pathologically confirmed to have lymph node metastasis after surgery. The study will proceed as follows:

Patients who have undergone cervical cancer surgery and have been pathologically confirmed to have positive retroperitoneal lymph nodes will be selected according to the inclusion and exclusion criteria. Their clinical and pathological data will be collected. These patients will be randomly assigned in a 1:1 ratio to two groups: the chemotherapy-immunotherapy (chemo-immunotherapy) group and the concurrent chemoradiotherapy group.

The study will compare the two treatment strategies by evaluating tumors' 3-year recurrence rate, distant metastasis rate, and overall survival prognosis in patients. The primary endpoints are the 3-year recurrence rate and distant metastasis rate. Secondary endpoints include the 3-year local recurrence rate, progression-free survival (PFS), and overall survival (OS). Additionally, the study will assess differences in complications, toxic side effects of chemotherapy and radiotherapy, and quality of life between the two groups to determine the value of chemo-immunotherapy in treating this patient population.

In addition, biological tissue samples from 50 patients in the chemo-immunotherapy cohort will be collected for multi-omics analysis and detection of immune-related biomarkers. Using bioinformatics methods, the study will analyze the differences in cellular immune subtypes and immune-related biomarkers between patients who benefit from the treatment and those who do not. This analysis aims to clarify the therapeutic efficacy of chemo-immunotherapy in patients with postoperative lymph node metastasis after cervical cancer surgery and to identify biomarkers and immune markers associated with treatment benefits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with cervical squamous cell carcinoma, adenocarcinoma (usual type), or adenosquamous carcinoma who have been pathologically confirmed to have positive retroperitoneal lymph nodes after radical surgery for cervical cancer, i.e., patients with stage IIIC1p and IIIC2p cervical cancer (FIGO 2018);
2. Positive expression of PD-L1 in pathological examination, i.e., Combined Positive Score (CPS) ≥1;
3. Patients aged ≥18 years and ≤70 years;
4. ECOG performance status score ≤1;
5. Laboratory tests: White blood cell count (WBC) ≥3.5×10^9/L, neutrophil count (NEU) ≥1.5×10^9/L, platelet count (PLT) ≥100×10^9/L, serum total bilirubin ≤1.5 times the upper limit of normal, serum alanine aminotransferase (ALT) and serum aspartate aminotransferase (AST) ≤1.5 times the upper limit of normal, serum blood urea nitrogen (BUN) ≤1.5 times the upper limit of regular or creatinine clearance rate ≥50 mL/min (creatinine clearance rate can be calculated using the Cockcroft-Gault formula, the Chronic Kidney Disease Epidemiology Collaboration formula, or the Modification of Diet in Renal Disease formula);
6. Good compliance of the subjects, who can follow the protocol for efficacy follow-up and adverse events/reactions;
7. Subjects voluntarily sign the informed consent form, including adherence to the requirements and restrictions listed in the informed consent form and this protocol.

Exclusion Criteria:

1. Postoperative pathology indicates positive parametrial involvement or positive surgical margins;
2. Incomplete radical surgery;
3. Postoperative imaging confirms the presence of residual target lesions;
4. Any active autoimmune disease or a history of autoimmune disease requiring systemic treatment, including but not limited to autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, thyroid dysfunction, and asthma requiring intervention with bronchodilators;
5. Previous treatment with immune checkpoint inhibitors, including but not limited to other anti-PD-1 and anti-PD-L1 antibodies; known allergy to any component of the study medication or other monoclonal antibodies;
6. History of human immunodeficiency virus (HIV) infection, active hepatitis B (HBV-DNA ≥ 2000 IU/mL or 10⁴ copies/mL), or hepatitis C (positive hepatitis C antibody and HCV-RNA above the lower limit of detection of the assay method);
7. Receipt of immunosuppressive drugs or systemic corticosteroid therapy for immunosuppressive purposes within 2 weeks before the study drug administration (dose >10 mg/day of prednisone or equivalent);
8. Diagnosis of another primary malignancy within 5 years before the first use of the investigational drug.
9. Use any other investigational drug/treatment from another clinical trial within 4 weeks before randomization or concurrent participation in another interventional clinical trial. Participation in observational, non-interventional clinical trials is permitted;
10. Pregnant or breastfeeding female patients;
11. Uncontrolled concomitant diseases, including but not limited to:

    * Cardiovascular diseases: New York Heart Association (NYHA) functional class II or higher, severe/unstable angina, myocardial infarction within ≤6 months before study drug administration, or significant arrhythmias requiring medication or intervention;
    * Uncontrolled hypertension;
    * Cerebrovascular events or central nervous system disorders within ≤6 months before study drug administration, or patients with abnormal mental status;
    * Hematologic disorders: Coagulopathy (INR > 2.0, PT > 16 seconds), bleeding tendency, or ongoing thrombolytic or anticoagulant therapy;
    * Hepatic or renal developmental abnormalities or history of surgery;
    * Any active infection requiring systemic antimicrobial therapy within 14 days before the first dose of the study drug;
12. Receipt of any live or attenuated vaccines within 4 weeks before the first dose of the study drug. Administration of seasonal inactivated influenza vaccine is permitted;
13. Patients who have previously undergone allogeneic bone marrow transplant or solid organ transplantation;
14. History of drug and/or alcohol abuse;
15. Patients deemed by the investigator unlikely to comply with study procedures, restrictions, and requirements are not eligible for participation in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year recurrence rate | From enrollment to the end of treatment at 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Womens' Hosptial, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No